CLINICAL TRIAL: NCT04862702
Title: Assessment of Postoperative Pain and Bacterial Load Reduction After Using TruNatomy and ProTaper Next Rotary Systems in Patients With Necrotic Mandibular Molars: A Randomized Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, yasmin hamdy hussien, Assitant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ENDO:3-3-5
Record Dates: First submitted 2020-10-14; First posted 2021-04-28 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Endodontic Treatment

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The assistant supervisor is the one who will generate the random sequence, assign the participants to the intervention or control groups and the only one who knows whether A or B represents the intervention or the control.
  The operators will enroll the participants after they find the eligible ones and confirm with the assistant supervisor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ProTaper Next rotary file system (Dentsply Sirona) (Active Comparator)
  Interventions: Device: mechanical instrumentation using rotary file system
- TruNatomy rotary system (Dentsply Sirona) (Experimental)
  Interventions: Device: mechanical instrumentation using rotary file system

INTERVENTIONS:
Device: mechanical instrumentation using rotary file system — the mechanical preparation will be performed using rotary file system

SUMMARY:
This study aims to assess the effect of rotary instrumentation using ProTaper Next rotary system versus TruNatomy rotary system on postoperative pain and the bacterial load reduction following single visit root canal treatment in necrotic mandibular molars.

DETAILED DESCRIPTION:
In the last years several rotary systems had launched to the market for mechanical preparation. The new era in the mechanical instrumentation aims to preserve the maximum amount of the peri-cervical dentine without affecting the proper cleaning and bacterial elimination. This will improve the long-term survival of the tooth with appropriate removal of microbes and microbial irritants.

ProTaper Next is a rotary system made from M wire. It is characterized by an innovative off-centered rectangular cross section that is suggested to give the files a snake-like swaggering movement as it advances into the root canal. This movement minimizes the engagement between the file and dentin and improves extruding debris out of the canal.

TruNatomy (Dentsply Sirona), is recently introduced as a new generation of rotary file system. TruNatomy files are designed to shape root canal systems to a continuously tapering preparation with maximum preservation of peri-cervical dentine. TruNatomy system offers a more safety, simplicity, improved cutting efficiency and mechanical properties compared to previous generations of rotating instruments, Many researches had been conducted to address the effect of ProTaper Next on post-operative pain considering it the most commonly used system. Thus, this study will be performed to evaluate and compare the influence of using the two systems on the intensity of postoperative pain and bacterial load reduction.

ELIGIBILITY:
Inclusion Criteria:

* - Medically free patients.
* Mandibular permanent molar teeth:
* Diagnosed clinically with pulp necrosis.
* Absence of spontaneous pain.
* Slight widening in the periodontal membrane space or with periapical radiolucency
* Patient's age ranges between 22 to 45 years with no sex predilection.
* Patients who can understand Modified Visual Analogue Scale (VAS).
* Patients' acceptance to participate in the trial.
* Patients able to sign informed consent.

Exclusion Criteria:

* - Medically compromised patients: Pain levels and healing following treatment would be compromised as these patients have shown higher incidence of pain and lower healing rate.
* Pregnant women: Avoid radiation exposure, anesthesia, and medication.
* If analgesics or antibiotics have been administrated by the patient during the past 24 hours preoperatively might alter their pain perception.
* Patients reporting bruxism or clenching: Avoid further pressure on an already inflamed tooth inducing subsequent irritation and inflammation.
* Teeth that show association with acute periapical abscess and swelling: Need special treatment steps which could involve additional visits with incision and drainage. Also, it could influence initiation and progression of postoperative pain.
* Greater than grade I mobility or pocket depth greater than 5mm. Need special surgical and/or periodontal therapy.
* No restorability: Hopeless tooth.
* Vital teeth.
* Immature teeth.
* Radiographic evidence of external or internal root resorption vertical root fracture, perforation, calcification.

Ages: 22 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Intensity of postoperative pain | 48 hours
  Postoperative pain will be measured by modified VAS at 6, 12, 24 and 48 hours post-obturation.
  The modified VAS consists of from 0-10 point scale anchored by two extremes "No pain" and "pain as bad as could be". The patients will be asked to choose the mark on an appendix that represents their level of pain. Pain level will be assigned to one of four categorical scores:
  1. None (0)
  2. Mild (1-3)
  3. Moderate (4-6)
  4. Severe (7-10) numerical rating scale (NRS) at 6, 12, 24 and 48 hours post-obturation and at 6, 12, 24 and 48 hours post-obturation.

SECONDARY OUTCOMES:
Bacterial load reduction | 24 hours
  Bacterial load reduction will be determined by bacterial counting using agar culture technique after root canal preparation (CFU/ml).

IPD SHARING:
Plan to Share IPD: Undecided